CLINICAL TRIAL: NCT00609102
Title: Antioxidant Treatment of Type 2 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: R. Paul Robertson, Pacific Northwest Research Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Antioxidant trmt type 2; NIH R01 38325-19
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- antioxidant drug (Active Comparator): n-acetylcysteine
  Interventions: Drug: n-aceylcysteine

INTERVENTIONS:
Drug: Placebo — one capsule BID
  Arms: Placebo
Drug: n-aceylcysteine — 450 mgm BID
  Arms: antioxidant drug

SUMMARY:
This study examines whether an antioxidant taken orally will improve glucose tolerance and insulin secretion in type 2 diabetic subjects.

ELIGIBILITY:
Inclusion Criteria: Subjects with a known diagnosis of type 2 diabetes -

Exclusion Criteria: None, except known intolerance to n-acetylcysteine

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 3 months

SECONDARY OUTCOMES:
HbA1c levels | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific Northwest Research Institute, Seattle, Washington, United States